CLINICAL TRIAL: NCT01106690
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Arm, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin and Pioglitazone Therapy
Brief Title: The CANTATA-MP Trial (CANagliflozin Treatment and Trial Analysis - Metformin and Pioglitazone)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017032; 28431754DIA3012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-01; First posted 2010-04-20 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Sitagliptin (Januvia); Metformin; Pioglitazone (Actos); Hemoglobin A1c; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo/Sitagliptin (Other): Each patient will receive matching placebo once daily for 26 weeks with stable doses of metformin and pioglitazone. At Week 26, patients will be switched from placebo to 100 mg of sitagliptin once daily with stable doses of metformin and pioglitazone until Week 52.
  Interventions: Drug: Placebo; Drug: Sitagliptin; Drug: Metformin; Drug: Pioglitazone
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone.
  Interventions: Drug: Canagliflozin; Drug: Metformin; Drug: Pioglitazone
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone.
  Interventions: Drug: Canagliflozin; Drug: Metformin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Placebo — One matching placebo capsule orally (by mouth) once daily for 26 weeks with stable doses of metformin and pioglitazone.
  Arms: Placebo/Sitagliptin
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally once daily for 52 weeks with stable doses of metformin and pioglitazone.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Sitagliptin — One 100 mg over-encapsulated tablet orally once daily beginning at Week 26 until Week 52 with stable doses of metformin and pioglitazone.
  Arms: Placebo/Sitagliptin
Drug: Metformin — The patient's stable dose of metformin background therapy should be continued throughout the study.
Drug: Pioglitazone — The patient's stable dose of pioglitazone background therapy should be continued throughout the study.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 different doses of canagliflozin compared with placebo in patients with type 2 diabetes mellitus who are receving treatment with metformin and pioglitazone and have inadequate glycemic (blood sugar) control.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (study drug assigned by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), parallel-group, 3-arm (3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of canagliflozin (100 mg and 300 mg) compared to placebo (a capsule that looks like all the other treatments but has no real medicine) in patients with T2DM who are not achieving an adequate response from current antihyperglycemic therapy with metformin and pioglitazone to control their diabetes. Approximately 360 patients with T2DM who are receiving combination therapy with metformin and pioglitazone will receive the addition of once-daily treatment with canagliflozin (100 mg or 300 mg) or placebo capsules for 26 weeks followed by a 26-week extension period where patients treated with canagliflozin (100 mg or 300 mg) will continue treatment for an additional 26 weeks and patients treated with placebo will be switched to active double-blind treatment with sitagliptin 100 mg, an antihyperglycemic agent administered once-daily for 26 weeks. In addition, all patients will take protocol specified stable doses of metformin and pioglitazone along with assigned study drug for the duration of the study. Patients will participate in the study for approximately 59 to 78 weeks. During the study, if a patient's fasting blood sugar remains high despite treatment with study drug, the patient will receive treatment with glimepiride (rescue therapy) in accordance with local prescribing information. During treatment, patients will be monitored for safety by review of adverse events, results from laboratory tests, 12-lead electrocardiograms (ECGs), vital signs measurements, body weight, physical examinations, and self-monitored blood glucose (SMGB) measurements. The primary outcome measure in the study is the effect of canagliflozin relative to placebo on hemoglobin A1c (HbA1c) after 26 weeks of treatment. Study drug will be taken orally (by mouth) once daily before the first meal each day unless otherwise specified. Patients will take single-blind placebo capsules for 2 weeks before randomization. After randomization, patients will take double-blind canagliflozin (100 mg or 300 mg) for 52 weeks OR placebo for 26 weeks switched to double-blind sitagliptin 100 mg for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM and be currently treated with PPAR gamma agent ((pioglitazone or rosiglitazone) and another anti-diabetes agent (metformin)
* Patients in the study must have a HbA1c between >=7 and <=10.5% and a fasting plasma glucose (FPG) <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* or a severe hypoglycemic episode within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (83):
- United States (41):
  - Anniston, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Burlingame, California
  - Encinitas, California
  - Fullerton, California
  - Roseville, California
  - Santa Ana, California
  - Wes Hills, California
  - Colorado Springs, Colorado
  - Bartow, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - Des Moines, Iowa
  - Baton Rouge, Louisiana
  - Chaska, Minnesota
  - Picayune, Mississippi
  - Billings, Montana
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Dublin, Ohio
  - Perrysburg, Ohio
  - Tulsa, Oklahoma
  - Yukon, Oklahoma
  - Bensalem, Pennsylvania
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Grand Prairie, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Virginia Beach, Virginia
  - Federal Way, Washington
  - Selah, Washington
- Canada (12):
  - Bathurst, New Brunswick
  - Moncton, New Brunswick
  - Grand Falls-Windsor, Newfoundland and Labrador
  - Brampton, Ontario
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Smiths Falls, Ontario
  - Thornhill, Ontario
  - Drummondville, Quebec
  - Calgary
  - Mount Pearl
  - Truro
- Finland (3):
  - Kuopio
  - Oulu
  - Turku
- France (3):
  - Bondy
  - Le Creusot
  - Narbonne
- Germany (4):
  - Aschaffenburg
  - Mainz
  - Neuwied
  - Schkeuditz
- Greece (3):
  - Athens
  - Thessaloniki
  - Thessalonikis
- India (6):
  - Ahmedabad
  - Belagavi
  - Chennai
  - Coimbatore
  - Jaipur
  - Nagpur
- Mexico (4):
  - Chihuahua City
  - Ciudad Juárez
  - Durango
  - México
- Spain (3):
  - Almería
  - Madrid
  - Seville
- Thailand (2):
  - Bangkok
  - Khon Kaen
- United Kingdom (2):
  - Antrim
  - Belfast

REFERENCES:
- [Derived] Davies MJ, Merton K, Vijapurkar U, Yee J, Qiu R. Efficacy and safety of canagliflozin in patients with type 2 diabetes based on history of cardiovascular disease or cardiovascular risk factors: a post hoc analysis of pooled data. Cardiovasc Diabetol. 2017 Mar 21;16(1):40. doi: 10.1186/s12933-017-0517-7. PMID 28327140
- [Derived] Pfeifer M, Townsend RR, Davies MJ, Vijapurkar U, Ren J. Effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on blood pressure and markers of arterial stiffness in patients with type 2 diabetes mellitus: a post hoc analysis. Cardiovasc Diabetol. 2017 Feb 27;16(1):29. doi: 10.1186/s12933-017-0511-0. PMID 28241822
- [Derived] Gilbert RE, Mende C, Vijapurkar U, Sha S, Davies MJ, Desai M. Effects of Canagliflozin on Serum Magnesium in Patients With Type 2 Diabetes Mellitus: A Post Hoc Analysis of Randomized Controlled Trials. Diabetes Ther. 2017 Apr;8(2):451-458. doi: 10.1007/s13300-017-0232-0. Epub 2017 Feb 14. PMID 28197834
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] John M, Cerdas S, Violante R, Deerochanawong C, Hassanein M, Slee A, Canovatchel W, Hamilton G. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus living in hot climates. Int J Clin Pract. 2016 Sep;70(9):775-85. doi: 10.1111/ijcp.12868. PMID 27600862
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Blonde L, Woo V, Mathieu C, Yee J, Vijapurkar U, Canovatchel W, Meininger G. Achievement of treatment goals with canagliflozin in patients with type 2 diabetes mellitus: a pooled analysis of randomized controlled trials. Curr Med Res Opin. 2015 Nov;31(11):1993-2000. doi: 10.1185/03007995.2015.1082991. Epub 2015 Sep 28. PMID 26373629
- [Derived] Gavin JR 3rd, Davies MJ, Davies M, Vijapurkar U, Alba M, Meininger G. The efficacy and safety of canagliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2015;31(9):1693-702. doi: 10.1185/03007995.2015.1067192. Epub 2015 Sep 4. PMID 26121561
- [Derived] Cefalu WT, Stenlof K, Leiter LA, Wilding JP, Blonde L, Polidori D, Xie J, Sullivan D, Usiskin K, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and relationship to HbA1c and blood pressure changes in patients with type 2 diabetes. Diabetologia. 2015 Jun;58(6):1183-7. doi: 10.1007/s00125-015-3547-2. Epub 2015 Mar 27. PMID 25813214
- [Derived] Weir MR, Januszewicz A, Gilbert RE, Vijapurkar U, Kline I, Fung A, Meininger G. Effect of canagliflozin on blood pressure and adverse events related to osmotic diuresis and reduced intravascular volume in patients with type 2 diabetes mellitus. J Clin Hypertens (Greenwich). 2014 Dec;16(12):875-82. doi: 10.1111/jch.12425. Epub 2014 Oct 20. PMID 25329038
- [Derived] Usiskin K, Kline I, Fung A, Mayer C, Meininger G. Safety and tolerability of canagliflozin in patients with type 2 diabetes mellitus: pooled analysis of phase 3 study results. Postgrad Med. 2014 May;126(3):16-34. doi: 10.3810/pgm.2014.05.2753. PMID 24918789
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Sinclair A, Bode B, Harris S, Vijapurkar U, Mayer C, Fung A, Shaw W, Usiskin K, Desai M, Meininger G. Efficacy and safety of canagliflozin compared with placebo in older patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. BMC Endocr Disord. 2014 Apr 18;14:37. doi: 10.1186/1472-6823-14-37. PMID 24742013
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus with inadequate control despite treatment with metformin and pioglitazone. The study was conducted between 13 April 2010 and 20 November 2011 and recruited patients from 74 study centers in 11 countries worldwide.
Pre-assignment Details: 344 patients were randomly allocated to the 3 treatment arms. 342 patients received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set (used for the Week 26 efficacy analysis) and safety analysis set (used for the Week 26 and Week 52 safety analyses).
Groups:
- Placebo/Sitagliptin: Each patient received matching placebo once daily for 26 weeks with stable doses of metformin and pioglitazone. At Week 26, patients were switched from placebo to 100 mg of sitagliptin once daily with stable doses of metformin and pioglitazone until Week 52.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone.
Period: Core Period: Baseline to Week 26
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 115 | 113 | 114
Completed | 91 | 104 | 101
Not Completed | 24 | 9 | 13
Not completed — Adverse Event | 6 | 1 | 4
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0
Not completed — Creatinine or eGFR withdrawal criteria | 0 | 3 | 1
Not completed — Noncompliance with study drug | 0 | 1 | 0
Not completed — Unable to take rescue therapy | 1 | 0 | 0
Not completed — Lack of efficacy on rescue therapy | 1 | 0 | 0
Not completed — Other | 10 | 2 | 6
Period: Extension Period: Week 26 to Week 52
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 90 (1 pt completed core but did not enter ext: physician decision(1).) | 103 (1 pt completed core but did not enter ext: physician decision(1).) | 96 (5 pts completed core but did not exter ext: lost to f/u(1), not spec(2), AE(1), eGFR criteria(1).)
Completed | 78 | 96 | 89
Not Completed | 12 | 7 | 7
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Noncompliance with study drug | 0 | 0 | 1
Not completed — Unable to take rescue therapy | 1 | 1 | 0
Not completed — Other | 8 | 3 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 115 | 113 | 114 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 83 | 83 | 83 | 249
  >=65 years | 32 | 30 | 31 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.56) | 56.7 (10.36) | 57 (10.19) | 57.4 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 51 | 126
  Male | 76 | 77 | 63 | 216
Region of Enrollment [Number; unit: participants]
  CANADA | 24 | 22 | 21 | 67
  FINLAND | 7 | 3 | 3 | 13
  FRANCE | 1 | 0 | 1 | 2
  GERMANY | 7 | 5 | 7 | 19
  GREECE | 0 | 0 | 1 | 1
  INDIA | 10 | 10 | 5 | 25
  MEXICO | 7 | 3 | 11 | 21
  SPAIN | 8 | 5 | 2 | 15
  THAILAND | 5 | 8 | 4 | 17
  UNITED KINGDOM | 3 | 2 | 3 | 8
  UNITED STATES | 43 | 55 | 56 | 154

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 114 | 113 | 112
Percent | -0.26 (0.069) | -0.89 (0.069) | -1.03 (0.070)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.62, 95% CI 2-sided [-0.811 to -0.437], Standard Error of Mean 0.095
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.76, 95% CI 2-sided [-0.951 to -0.575], Standard Error of Mean 0.096

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26
Description: The table below shows the percentage of patients with HbA1c<7% at Week 26 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 114 | 113 | 112
Percentage of patients | 32.5 | 46.9 | 64.3
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.40, 95% CI [1.26 to 4.57]
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.38, 95% CI 2-sided [2.73 to 10.60]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 114 | 113 | 112
mg/dL | 2.54 (2.785) | -26.8 (2.796) | -33.2 (2.817)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -29.4, 95% CI 2-sided [-36.96 to -21.78], Standard Error of Mean 3.857
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -35.7, 95% CI 2-sided [-43.30 to -28.11], Standard Error of Mean 3.861

4. Secondary Outcome: Change in Homeostasis Model Assessment (HOMA2-%B) From Baseline to Week 26
Description: HOMA2-%B is a measure of beta cell function (the cells in the pancreas that produce and store insulin). The table below shows the least-squares (LS) mean change in HOMA2-%B from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: HOMA2-%B
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 100 | 103 | 105
HOMA2-%B | 0.91 (1.833) | 15.19 (1.809) | 18.14 (1.790)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 14.28, 95% CI 2-sided [9.315 to 19.236], Standard Error of Mean 2.521
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 17.23, 95% CI 2-sided [12.293 to 22.166], Standard Error of Mean 2.509

5. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 114 | 113 | 112
Percent change | -0.1 (0.3) | -2.8 (0.3) | -3.8 (0.3)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -2.7, 95% CI 2-sided [-3.6 to -1.8], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -3.7, 95% CI 2-sided [-4.6 to -2.8], Standard Error of Mean 0.4

6. Secondary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in SBP from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 114 | 113 | 112
mmHg | -1.24 (1.033) | -5.30 (1.036) | -4.70 (1.044)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; Least-Squares Mean Difference = -4.07, 95% CI 2-sided [-6.879 to -1.251], Standard Error of Mean 1.430
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.016, ANCOVA; Least-Squares Mean Difference = -3.46, 95% CI 2-sided [-6.281 to -0.643], Standard Error of Mean 1.433

7. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in triglycerides from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 105 | 108 | 109
Percent change | 15.2 (4.1) | 3.2 (4.1) | -1.7 (4.1)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.034, ANCOVA; Least-Squares Mean Difference = -12.1, 95% CI 2-sided [-12.1 to -0.9], Standard Error of Mean 5.7
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; Least-Squares Mean Difference = -16.9, 95% CI 2-sided [-28.1 to -5.8], Standard Error of Mean 5.7

8. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean percent change in HDL-C from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo/Sitagliptin | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 105 | 107 | 109
Percent change | 2.4 (1.4) | 7.2 (1.3) | 8.9 (1.3)
Statistical Analysis 1: Comparison: Placebo/Sitagliptin vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.010, ANCOVA; Least-Squares Mean Difference = 4.8, 95% CI 2-sided [1.2 to 8.5], Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: Placebo/Sitagliptin vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = 6.5, 95% CI 2-sided [2.8 to 10.2], Standard Error of Mean 1.9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of study (52 weeks).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm either during the 26-week period or entire 52-week period.
Groups:
- Placebo/Sitagliptin: Baseline to Week 26: Each patient received matching placebo once daily for 26 weeks with stable doses of metformin and pioglitazone. At Week 26, patients were switched from placebo to 100 mg of sitagliptin once daily with stable doses of metformin and pioglitazone until Week 52. Data are presented for Baseline to Week 26.
- Canagliflozin 100 mg: Baseline to Week 26: Each patient received 100 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone. Data are presented for Baseline to Week 26.
- Canagliflozin 300 mg: Baseline to Week 26: Each patient received 300 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone. Data are presented for Baseline to Week 26.
- Placebo/Sitagliptin: Baseline to Week 52: Each patient received matching placebo once daily for 26 weeks with stable doses of metformin and pioglitazone. At Week 26, patients were switched from placebo to 100 mg of sitagliptin once daily with stable doses of metformin and pioglitazone until Week 52. Data are presented for Baseline to Week 52.
- Canagliflozin 100 mg: Baseline to Week 52: Each patient received 100 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone. Data are presented for Baseline to Week 52.
- Canagliflozin 300 mg: Baseline to Week 52: Each patient received 300 mg of canagliflozin once daily for 52 weeks with stable doses of metformin and pioglitazone. Data are presented for Baseline to Week 52.
Arm/Group | Placebo/Sitagliptin: Baseline to Week 26 | Canagliflozin 100 mg: Baseline to Week 26 | Canagliflozin 300 mg: Baseline to Week 26 | Placebo/Sitagliptin: Baseline to Week 52 | Canagliflozin 100 mg: Baseline to Week 52 | Canagliflozin 300 mg: Baseline to Week 52
Serious Adverse Events (participants affected / at risk) | 5/115 | 3/113 | 4/114 | 6/115 | 8/113 | 7/114
Other Adverse Events (participants affected / at risk) | 31/115 | 35/113 | 40/114 | 49/115 | 48/113 | 57/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sitagliptin: Baseline to Week 26 (N=115) | Canagliflozin 100 mg: Baseline to Week 26 (N=113) | Canagliflozin 300 mg: Baseline to Week 26 (N=114) | Placebo/Sitagliptin: Baseline to Week 52 (N=115) | Canagliflozin 100 mg: Baseline to Week 52 (N=113) | Canagliflozin 300 mg: Baseline to Week 52 (N=114)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52.
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Arteriogram coronary (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sitagliptin: Baseline to Week 26 (N=115) | Canagliflozin 100 mg: Baseline to Week 26 (N=113) | Canagliflozin 300 mg: Baseline to Week 26 (N=114) | Placebo/Sitagliptin: Baseline to Week 52 (N=115) | Canagliflozin 100 mg: Baseline to Week 52 (N=113) | Canagliflozin 300 mg: Baseline to Week 52 (N=114)
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 4 | 7 | 7 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Nasopharyngitis (Infections and infestations) | 6 | 6 | 11 | 13 | 11 | 15 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Upper respiratory tract infection (Infections and infestations) | 7 | 9 | 5 | 9 | 14 | 8 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Urinary tract infection (Infections and infestations) | 6 | 4 | 4 | 9 | 5 | 9 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 3 | 6 | 1 | 3 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 6 | 3 | 3 | 5 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52. In the Week 26 study report, 2 patients had hypoglycaemia recorded in error by the investigator, which were corrected in the Week 52 study report.
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 3 | 3 | 9 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5 | 4 | 10 | 7 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Pollakiuria (Renal and urinary disorders) | 1 | 5 | 7 | 1 | 6 | 8 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1 | 7 | 5 | 2 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Oedema peripheral (General disorders) | 2 | 2 | 4 | 4 | 2 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52.
Headache (Nervous system disorders) | 4 | 3 | 5 | 5 | 3 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52.
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 6 | 2 | 4 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.